CLINICAL TRIAL: NCT01391923
Title: Non-Invasive Reduction of Fat in the Arms With the CoolFlex Applicator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA11-002
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2012-03

CONDITIONS: Fat Reduction in the Upper Arm
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study is being performed to reduce unwanted fat in the arm using a new applicator for the Zeltiq System.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and performance of the CoolFlex applicator in the flat configuration for reduction of fat in the upper arms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on the underside of the upper arm, generally located over the triceps muscle. (Figure 1)
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject agrees to maintain their weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
5. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction or mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
4. Subject needs to administer, or has a known history of, subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject body mass index (BMI) exceeds 40. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
9. Subject is taking or has taken diet pills or supplements within the past month.
10. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation.
11. Subject is pregnant or intending to become pregnant in the next 6 months.
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject is unable or unwilling to comply with the study requirements.
14. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Independent imaging review | 16 weeks
  Performance will be evaluated by changes in the contour as established by blinded photographic review of a series of pre- and 16-week post-treatment images for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Boey, MD, Principal Investigator — Arbutus Laser Centre
Locations (2):
- Canada (2):
  - Arbutus Laser Centre, Vancouver, British Columbia
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario

IPD SHARING:
Plan to Share IPD: No